CLINICAL TRIAL: NCT05370742
Title: Comparison of Clinical and Radiological Results of Using Only Screws and Plate Use in Latarjet Operation in Shoulder Instability
Status: Temporarily not available | Type: Expanded Access
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, oguzhan albayrak, medical doctor, Istanbul University
Other Study IDs: oalbayrak
Record Dates: First submitted 2022-04-28; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Bone Plates

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Procedure: Latarjet surgery — Results of using a screw-only plate for fixation of the corocoid bone in recurrent shoulder dislocations
  Other Names: smith and nephew brand screws and plates

SUMMARY:
Randomized controlled comparison of the clinical and radiological results of using only screws and plate use in latarjet surgery in shoulder instability

DETAILED DESCRIPTION:
Randomized controlled comparison of the clinical and radiological results of using only screws and plate use in latarjet surgery in shoulder instability

2 groups will be determined in the study, while the first group will include the group in which corocoid fixation with cannulated screws was performed, while the second group will include the group that underwent osteosynthesis with plate and screw

The results will be evaluated statistically based on clinical scores (constant, vas) and radiological findings (a angle).

ELIGIBILITY:
Inclusion Criteria:

- Recurrent shoulder dislocation; 18-65 age

>%10 glenoid loss or Hill Sacs Lesion

Exclusion Criteria:

- <18 age <%10 glenoid loss shoulder dislocation due to epilepsy Dislocations associated with other upper extremity injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — a similar number of men and women will be selected

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Unıversıty faculty of medicine, Istanbul, Fatih/Topkapı, Turkey (Türkiye)